CLINICAL TRIAL: NCT01434563
Title: The CNS HAND Study: The Prevalence of Neurocognitive Disorder in a Primary Care-based HIV Cohort Compared to a HIV-negative Control Cohort
Brief Title: The Prevalence of Neurocognitive Disorder in a Primary Care-based HIV Cohort Compared to a HIV-negative Control Cohort -
Acronym: CNS HAND
Status: Completed | Type: Observational
Sponsor: Holdsworth House Medical Practice (Other)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Doctor, Holdsworth House Medical Practice
Other Study IDs: CNS HAND Study
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: HIV-1-Associated Cognitive Motor Complex
Keywords: HIV; neurocognitive disorder; primary care; HIV negative; HAND; CNS
MeSH Terms: conditions — AIDS Dementia Complex; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV positive: Subjects must have documented HIV, be english speaking, with life expectancy greater than 6 months, and must have adequate information available in their medical record to apply HAND predictive algorithm (HIV-associated neurological disease)
- HIV negative: Must have documented negative HIV test within 12 months of study entry, have no traumatic brain injury or history of chronic neurological illness/psychiatric conditions (such as bipolar or depression),be english speaking and have no history of drug or alcohol abuse.

SUMMARY:
To determine the prevalence of HIV associated Neurological Disorder (HAND) in a population of HIV positive patients within a primary care setting compared with the HIV negative population. The investigators aim is to assess the use of optimal screening methods to assess HAND. For this the investigators will be comparing the performance of a group of persons who are HIV positive and a group of persons who are HIV negative to test their memory and concentration abilities over-time.

ELIGIBILITY:
HIV positive Inclusion Criteria:

* Documented HIV infection
* Able to participate in study procedures

HIV positive Exclusion Criteria:

* Inability to comprehend or read English (as established by the English proficiency questionnaire)
* Drug or alcohol intoxicated (as determined by the investigator)
* Lack of information in medical records to determine the HAND predictive algorithm (current CD4 count, past CNS HIV-related disease, and duration of HIV therapy)
* Life expectancy <6 months
* Inability to attend the clinic for required study follow up visits

HIV-negative Inclusion Criteria:

* Negative HIV-1 test within 12 months of study entry

HIV-negative Exclusion Criteria:

* Life time traumatic brain injury leading to loss of consciousness of at least 30 minutes.
* Inability to comprehend or read English (as established by the English proficiency questionnaire).
* Inability to attend the clinic for required study follow up visits.
* History of chronic neurological illness.
* Unstable psychiatric conditions such as bipolar disorder or depression.
* Individuals with psychiatric disorder on the psychotic axis.
* Active or past (within the last 6 months) severe alcohol or substance abuse sufficient, in the investigator's judgement, to prevent completion of tests or Inability to attend for the planned required study follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending Holdsworth House Medical Practice, Sydney, Australia
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is percentage of patients with abnormal (-1.5 SD in 2 domains) CogState battery in HIV positive patients vs HIV negative patients. | 12 months
  The primary outcome measure is percentage of patients with abnormal (-1.5 SD in 2 domains) CogState battery in HIV positive patients vs HIV negative patients.